CLINICAL TRIAL: NCT01723787
Title: Genetic Studies in Patients and Families With Infantile Spasms
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 12-0482
Record Dates: First submitted 2012-11-06; First posted 2012-11-08 (Estimated); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Infantile Spasms
MeSH Terms: conditions — Spasms, Infantile

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, saliva, buccal cells,urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Infantile Spasms: Participants retrospectively identified to have been treated with ACTH according to FDA-approved protocol for Infantile Spasms
- biological parents: Biological parents of participants retrospectively identified to have been treated with ACTH according to FDA-approved protocol for Infantile Spasms

SUMMARY:
Infantile spasms (IIS), a characteristic epilepsy syndrome of infancy with often catastrophic developmental consequences, is known in some patients to have many different genetic, metabolic and structural etiologies. However, for most patients IIS is the only presenting clinical feature and the specific cause is unknown. Only two FDA approved pharmacologic treatments for IIS exist, Adrenocorticotropic hormone (ACTH) and vigabatrin. While vigabatrin may be the treatment of choice for Tuberous Sclerosis as a cause for IS, ACTH is the treatment of choice for all others. Unfortunately, a substantial number of patients may still not respond to ACTH and there is no a priori way that suggests which patients may be responders. This has led to the following key questions:

Can novel genetic analyses determine known genetic causes of IS with greater efficiency (more timely and cost-effective)? Can novel genetic analyses determine previously unknown disease modifying genes that predispose individuals to develop IS? Can novel genetic analyses elaborate genes and gene polymorphisms that favor ACTH responsiveness? Do these polymorphisms suggest strategies to improve ACTH responsiveness?

DETAILED DESCRIPTION:
Primary Aim 1: Apply whole-exome sequencing to determine possible causes of cryptogenic IS and evaluate adding whole-exome sequencing to standard practice for determining causes of IS. Sub-aim 1: Determine the effectiveness of whole-exome sequencing in suggesting disease-modifying genes that may contribute to triggering IS.

Primary Aim 2: Determine genes, through whole-exome sequencing, that may play a role in determining ACTH responsiveness for IS. Sub-aim 2: Correlate genes or genetic factors (haplotypes) associated with ACTH responsiveness and disease modification.

ELIGIBILITY:
Inclusion Criteria:

* Patient trios (both biological parents + patient with IIS = trio) with IIS retrospectively identified to have been treated with ACTH according to FDA-approved protocol (Table 1).
* Ability to provide informed consent (in case of severe to profound intellectual disability, consent provided by an legally authorized representative, as necessary)

Exclusion Criteria:

* IIS due to suspected or genetically proven tuberous sclerosis
* IIS but do not meet retrospective enrollment criteria (Table 1)
* Inability to complete consent process

Ages: 31 Days to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All patients trios (both parents + patient with IIS = trio) with IIS retrospectively identified to have been treated with ACTH according to FDA-approved protocol will be eligible for inclusion in this study regardless of age, sex, ethnicity/race, or socioeconomic status. The principal recruitment venues will be Neurology clinics, in-patient service and Medical Genetics Clinics at Children's Hospital Colorado and University of Colorado Health Sciences Center (UCHSC)
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2013-03; Primary Completion 2017-03-09 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Determine the effectiveness of novel genetic analyses in suggesting disease-modifying genes that may contribute to triggering IIS. | Results of the DNA studies will be evaluated prior to completion of the 5th year to assess the need for further investigations.
  Apply novel genetic analyses to determine possible causes of cryptogenic IIS and evaluate adding novel genetic analyses to standard practice for determining causes of IIS

SECONDARY OUTCOMES:
Determine genes, through novel genetic analyses, that may play a role in determining ACTH responsiveness for IIS | Results of the DNA studies will be evaluated prior to completion of the 5th year to assess the need for further investigations
  Correlate genes or genetic factors (haplotypes) associated with ACTH responsiveness and disease modification

CONTACTS AND LOCATIONS:
Overall Officials: Tim Benke, MD, Principal Investigator — Children's Hospital Colorado
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States